CLINICAL TRIAL: NCT02113241
Title: Effect of Dapagliflozin Administration on Metabolic Syndrome, Insulin Sensitivity, and Insulin Secretion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Senior Researcher, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAPA-MS
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Metabolic Syndrome X
Keywords: metabolic syndrome; forxiga; dapagliflozin; insulin secretion; insulin sensitivity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin capsules, 10 mg, one per day before breakfast during 90 days.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo capsules, 10 mg, one per day before breakfast during 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin capsules, 10 mg, one per day before breakfast during 90 days.
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo — Placebo capsules, 10 mg, one per day before breakfast during 90 days.
  Other Names: Calcined magnesium
  Arms: Placebo

SUMMARY:
The Metabolic Syndrome is a high prevalence disease worldwide. About a quarter of the adult population suffers the disease.

Dapagliflozin is an inhibitor of the sodium-glucose co-transporter SGLT2 in the kidney and is a novel treatment for diabetes type 2. Some studies indicate that SGLT2 inhibitors have benefits on blood pressure, triglycerides levels and help to raise the levels of high density lipoproteins cholesterol (c-HDL).

The aim of this study is to evaluate the effect of dapagliflozin on metabolic syndrome, insulin sensitivity and insulin secretion.

The investigators hypothesis is that the administration of dapagliflozin modifies the metabolic syndrome, insulin sensitivity and insulin secretion.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial its going to carry out in 24 patients with a diagnosis of metabolic syndrome in accordance with the International Diabetes Federation (IDF). Waist circumference, glucose, insulin levels, lipid profile, creatinine and acid uric are going to be load after a 75 g of dextrose load.

12 patients will receive Forxiga (dapagliflozin), 10 mg, one per day before breakfast during 3 months.

The remaining 12 patients will receive placebo at the same dose.

There will be calculated Area Under the Curve of glucose and insulin, total insulin secretion (insulinogenic index), first-phase of insulin secretion (Stumvoll index) and insulin sensitivity (Matsuda index).

This protocol it's already approved by the local ethics committee and written informed consent it's going to be obtained from all volunteers.

Results will be presented as mean and standard deviation. Intra and inter group differences are going to be tested using the Wilcoxon signed-rank and Mann-Whitney U-test respectively; p≤0.05 it's going to be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 30 and 60 years
* Metabolic Syndrome according to the IDF criteria
* Waist circumference
* Man ≥90 cm
* Woman ≥80 cm
* And two of the following criteria
* High density lipoprotein
* Man ≤40 mg/dL
* Woman ≤50 mg/dL
* Fasting glucose ≥100 mg/dL
* Triglycerides ≥150 mg/dL
* Blood pressure ≥130/85 mmHg
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to SGLT2 inhibitors
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Previous treatment for the metabolic syndrome components
* Body Mass Index ≥39.9 kg/m2
* Fasting glucose ≥126 mg/dL
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥240 mg/dL
* Low density lipoprotein (c-LDL) ≥190 mg/dL
* Blood Pressure ≥140/90 mmHg

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Bolinder J, Ljunggren O, Kullberg J, Johansson L, Wilding J, Langkilde AM, Sugg J, Parikh S. Effects of dapagliflozin on body weight, total fat mass, and regional adipose tissue distribution in patients with type 2 diabetes mellitus with inadequate glycemic control on metformin. J Clin Endocrinol Metab. 2012 Mar;97(3):1020-31. doi: 10.1210/jc.2011-2260. Epub 2012 Jan 11. PMID 22238392
- [Background] Rosenstock J, Vico M, Wei L, Salsali A, List JF. Effects of dapagliflozin, an SGLT2 inhibitor, on HbA(1c), body weight, and hypoglycemia risk in patients with type 2 diabetes inadequately controlled on pioglitazone monotherapy. Diabetes Care. 2012 Jul;35(7):1473-8. doi: 10.2337/dc11-1693. Epub 2012 Mar 23. PMID 22446170
- [Background] Chao EC. Dapagliflozin: an evidence-based review of its potential in the treatment of type-2 diabetes. Core Evid. 2012;7:21-8. doi: 10.2147/CE.S16359. Epub 2012 Jun 1. PMID 22701099
- [Background] Kasichayanula S, Liu X, Lacreta F, Griffen SC, Boulton DW. Clinical pharmacokinetics and pharmacodynamics of dapagliflozin, a selective inhibitor of sodium-glucose co-transporter type 2. Clin Pharmacokinet. 2014 Jan;53(1):17-27. doi: 10.1007/s40262-013-0104-3. PMID 24105299
- [Background] Yang L, Li H, Li H, Bui A, Chang M, Liu X, Kasichayanula S, Griffen SC, Lacreta FP, Boulton DW. Pharmacokinetic and pharmacodynamic properties of single- and multiple-dose of dapagliflozin, a selective inhibitor of SGLT2, in healthy Chinese subjects. Clin Ther. 2013 Aug;35(8):1211-1222.e2. doi: 10.1016/j.clinthera.2013.06.017. Epub 2013 Aug 2. PMID 23910664
- [Background] Obermeier M, Yao M, Khanna A, Koplowitz B, Zhu M, Li W, Komoroski B, Kasichayanula S, Discenza L, Washburn W, Meng W, Ellsworth BA, Whaley JM, Humphreys WG. In vitro characterization and pharmacokinetics of dapagliflozin (BMS-512148), a potent sodium-glucose cotransporter type II inhibitor, in animals and humans. Drug Metab Dispos. 2010 Mar;38(3):405-14. doi: 10.1124/dmd.109.029165. Epub 2009 Dec 8. PMID 19996149
- [Background] Kasichayanula S, Liu X, Pe Benito M, Yao M, Pfister M, LaCreta FP, Humphreys WG, Boulton DW. The influence of kidney function on dapagliflozin exposure, metabolism and pharmacodynamics in healthy subjects and in patients with type 2 diabetes mellitus. Br J Clin Pharmacol. 2013 Sep;76(3):432-44. doi: 10.1111/bcp.12056. PMID 23210765
- [Background] Kilov G, Leow S, Thomas M. SGLT2 inhibition with dapagliflozin -- a novel approach for the management of type 2 diabetes. Aust Fam Physician. 2013 Oct;42(10):706-10. PMID 24130972
- [Background] Kaku K, Inoue S, Matsuoka O, Kiyosue A, Azuma H, Hayashi N, Tokudome T, Langkilde AM, Parikh S. Efficacy and safety of dapagliflozin as a monotherapy for type 2 diabetes mellitus in Japanese patients with inadequate glycaemic control: a phase II multicentre, randomized, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2013 May;15(5):432-40. doi: 10.1111/dom.12047. Epub 2013 Jan 25. PMID 23194084
- [Background] Zhang L, Feng Y, List J, Kasichayanula S, Pfister M. Dapagliflozin treatment in patients with different stages of type 2 diabetes mellitus: effects on glycaemic control and body weight. Diabetes Obes Metab. 2010 Jun;12(6):510-6. doi: 10.1111/j.1463-1326.2010.01216.x. PMID 20518806
- [Background] Lambers Heerspink HJ, de Zeeuw D, Wie L, Leslie B, List J. Dapagliflozin a glucose-regulating drug with diuretic properties in subjects with type 2 diabetes. Diabetes Obes Metab. 2013 Sep;15(9):853-62. doi: 10.1111/dom.12127. Epub 2013 Jun 5. PMID 23668478
- [Background] Ferrannini E, Ramos SJ, Salsali A, Tang W, List JF. Dapagliflozin monotherapy in type 2 diabetic patients with inadequate glycemic control by diet and exercise: a randomized, double-blind, placebo-controlled, phase 3 trial. Diabetes Care. 2010 Oct;33(10):2217-24. doi: 10.2337/dc10-0612. Epub 2010 Jun 21. PMID 20566676
- [Background] Bolinder J, Ljunggren O, Johansson L, Wilding J, Langkilde AM, Sjostrom CD, Sugg J, Parikh S. Dapagliflozin maintains glycaemic control while reducing weight and body fat mass over 2 years in patients with type 2 diabetes mellitus inadequately controlled on metformin. Diabetes Obes Metab. 2014 Feb;16(2):159-69. doi: 10.1111/dom.12189. Epub 2013 Aug 29. PMID 23906445
- [Background] Merovci A, Solis-Herrera C, Daniele G, Eldor R, Fiorentino TV, Tripathy D, Xiong J, Perez Z, Norton L, Abdul-Ghani MA, DeFronzo RA. Dapagliflozin improves muscle insulin sensitivity but enhances endogenous glucose production. J Clin Invest. 2014 Feb;124(2):509-14. doi: 10.1172/JCI70704. Epub 2014 Jan 27. PMID 24463448

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (8.4) | 49.5 (6.0) | 46.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Body weight (kg) [Mean (Standard Deviation); unit: kilograms] | 82.7 (12.9) | 80.0 (11.3) | 81.4 (12.0)
Body Mass Index (BMI) (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 33.3 (3.5) | 31.5 (3.1) | 32.5 (3.4)
Fat mass (kg) [Mean (Standard Deviation); unit: kilograms] | 33.2 (8.5) | 32.6 (8.2) | 32.9 (8.2)
Waist circumference (WC) (cm) [Mean (Standard Deviation); unit: centimeters] | 101.5 (10.1) | 96.1 (7.2) | 98.9 (9.1)
Systolic Blood Pressure (SBP) (mmHg) [Mean (Standard Deviation); unit: mmHg] | 121 (13) | 126 (10) | 123.8 (11.9)
Diastolic Blood Pressure (DBP) (mmHg) [Mean (Standard Deviation); unit: mmHg] | 78 (12) | 79 (10) | 78.2 (11.7)
Glucose at minute 0 (0') (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal (minute 0') and at the minutes 30 (30'), 60 (60'), 90 (90') and 120 (120') after a 75 g oral dextrose load.
  mmol/L | 6.1 (0.5) | 5.8 (0.6) | 6.0 (0.6)
Glucose at minute 30 (30') (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal (minute 0') and at the minutes 30 (30'), 60 (60'), 90 (90') and 120 (120') after a 75 g oral dextrose load.
  mmol/L | 10.7 (2.6) | 9.1 (2.1) | 9.9 (2.4)
Glucose at minute 60 (60') (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal (minute 0') and at the minutes 30 (30'), 60 (60'), 90 (90') and 120 (120') after a 75 g oral dextrose load.
  mmol/L | 12.0 (3.8) | 10.4 (2.6) | 11.2 (3.3)
Glucose at minute 90 (90') (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal (minute 0') and at the minutes 30 (30'), 60 (60'), 90 (90') and 120 (120') after a 75 g oral dextrose load.
  mmol/L | 10.9 (3.1) | 9.1 (2.6) | 10.0 (2.9)
Glucose at minute 120 (120') (mmol/L) [Mean (Standard Deviation); unit: mmol/L] — The blood samples were taken after the insertion of a catheter as an open path to facilitate the procedure. Blood samples were taken at the basal (minute 0') and at the minutes 30 (30'), 60 (60'), 90 (90') and 120 (120') after a 75 g oral dextrose load.
  mmol/L | 8.9 (2.1) | 7.6 (2.2) | 8.3 (2.2)
Total cholesterol (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 5.4 (0.7) | 4.9 (1.0) | 5.2 (0.9)
Triglycerides (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 2.7 (1.4) | 2.0 (0.7) | 2.4 (1.2)
HDL-cholesterol (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 1.2 (0.2) | 1.2 (0.3) | 1.2 (0.3)
LDL-cholesterol (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 2.9 (1.0) | 2.8 (0.9) | 2.9 (1.0)
Area Under the Curve (AUC) glucose (mmol*hr/L) [Mean (Standard Deviation); unit: mmol*hr/L] | 1235 (304) | 1060 (233) | 1148.3 (280)
Area Under the Curve (AUC) insulin (pmol*hr/L) [Mean (Standard Deviation); unit: pmol*hr/L] | 103910 (55167) | 106683 (41787) | 105297 (47884)
Insulinogenic index (total insulin secretion) [Mean (Standard Deviation); unit: index] — The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔAUC insulin/ΔAUC glucose), the entered values reflect the total insulin secretion
  index | 0.83 (0.64) | 0.98 (0.46) | 0.91 (0.55)
Stumvoll Index (first phase of insulin secretion) [Mean (Standard Deviation); unit: index] — Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
  index | 1566 (1137) | 1675 (819) | 1620.8 (971)
Matsuda Index (insulin sensitivity) [Mean (Standard Deviation); unit: index] — Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
  index | 2.0 (1.1) | 1.8 (0.8) | 1.9 (1.0)
Creatinine (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 0.06 (0.02) | 0.07 (0.02) | 0.07 (0.02)
Uric acid (umol/L) [Mean (Standard Deviation); unit: umol/L] | 267.7 (95.2) | 315.2 (101.1) | 291.5 (101.1)
Alanine aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] | 50.9 (31.6) | 37.9 (17.1) | 44.4 (25.7)
Aspartate aminotransferase (AST) [Mean (Standard Deviation); unit: U/L] | 37.9 (19.1) | 28.8 (17.7) | 33.4 (18.6)

OUTCOME MEASURES:

1. Primary Outcome: Waist Circumference at Week 12.
Description: The waist circumference is going to be evaluated at week 12 with a flexible tape with standardized techniques.
Time Frame: Week 12
Population: All participants, including those who dropped out before the end were taken into account for statistical analysis (intention to treat)
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
centimeters | 97.6 (8.9) | 97.2 (6.9)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.089, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

2. Primary Outcome: Triglycerides Levels at Week 12.
Description: The triglycerides levels are going to be evaluated at week 12 with enzymatic-colorimetric techniques.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 1.7 (0.8) | 1.7 (0.6)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.248, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

3. Primary Outcome: High Density Lipoprotein (c-HDL) Levels at Week 12.
Description: The c-HDL levels are going to be evaluated at week 12 with enzymatic/colorimetric techniques.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 1.3 (0.2) | 1.3 (0.2)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.161, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.079, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

4. Primary Outcome: Glucose Levels at Minute 0 at Week 12.
Description: The fasting glucose (0') levels are going to be evaluated at week 12 with enzymatic/colorimetric techniques.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 5.7 (1.1) | 5.8 (0.7)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.067, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.918, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

5. Primary Outcome: Systolic Blood Pressure at Week 12.
Description: The systolic blood pressure is going to be evaluated at week 12 with a digital sphygmomanometer.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmHg | 117 (10) | 121 (13)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.128, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.454, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

6. Primary Outcome: Diastolic Blood Pressure at Week 12.
Description: The diastolic blood pressure is going to be evaluated at week 12 with a digital sphygmomanometer.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmHg | 76 (8) | 79 (10)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.433, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.407, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

7. Primary Outcome: Insulinogenic Index (Total Insulin Secretion) at Week 12.
Description: The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔAUC insulin/ΔAUC glucose), the entered values reflect the total insulin secretion at week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
index | 0.35 (0.11) | 0.99 (0.38)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.826, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

8. Primary Outcome: Stumvoll Index (First Phase of Insulin Secretion) at Week 12.
Description: Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the frst phase of insulin secretion at week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
index | 1463 (879) | 2198 (996)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.791, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.413, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

9. Primary Outcome: Matsuda Index (Total Insulin Sensitivity) at Week 12.
Description: Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity at week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
index | 2.7 (1.4) | 1.6 (0.8)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.075, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.432, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

10. Secondary Outcome: Body Weight at Week 12.
Description: The weight it's going to be measured at week 12 with a bioimpedance balance.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
kilograms | 81.2 (12.8) | 79.6 (11.3)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.835, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

11. Secondary Outcome: Body Mass Index at Week 12
Description: The Body Mass index it's going to be calculated at week 12 with the Quetelet index.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
kg/m^2 | 32.6 (3.6) | 32.1 (2.7)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.778, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

12. Secondary Outcome: Fat Mass at Week 12.
Description: The fat mass is going to be evaluated at week 12 through bioimpedance.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
kilograms | 32.7 (9.2) | 34.4 (7.3)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.338, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.309, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

13. Secondary Outcome: Total Cholesterol at Week 12
Description: The total cholesterol will be estimated by standardized techniques at week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 5.2 (0.7) | 4.9 (0.8)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.049, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.563, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

14. Secondary Outcome: Low Density Lipoproteins (c-LDL) at Week 12
Description: The c-LDL levels are going to be measured at week 12 with standardized techniques.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 3.1 (0.5) | 2.8 (0.9)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.850, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.206, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

15. Secondary Outcome: Alanine Aminotransferase (ALT) at Week 12.
Description: The ALT hepatic transaminase levels are going to be measured at week 12 with standardized techniques.
Time Frame: Week 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
U/L | 32.1 (15.9) | 38.1 (25.0)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.950, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

16. Secondary Outcome: Aspartate Aminotransferase (AST) at Week 12.
Description: The hepatic transaminase AST will be evaluated with standardized methods at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
U/L | 31.1 (14.5) | 29.5 (16.5)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.011, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.454, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

17. Secondary Outcome: Creatinine at Week 12.
Description: The creatinine levels are going to be measured at week 12 with standardized techniques.
Time Frame: Week 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 0.07 (0.01) | 0.05 (0.02)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.652, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.055, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

18. Secondary Outcome: Uric Acid at Week 12.
Description: The uric acid levels are going to be measured at week 12 with standardized techniques.
Time Frame: Week 12.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
umol/L | 243.9 (55.3) | 339.0 (53.5)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.254, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.787, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

19. Secondary Outcome: AUC of Glucose at Week 12.
Description: The AUC of glucose will be calculated from the glucose values obtained from the minuted oral glucose tolerance curve at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol*hr/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol*hr/L | 1153 (280) | 1129 (232)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.129, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.365, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

20. Secondary Outcome: AUC of Insulin at Week 12.
Description: The AUC will be calculated from the insulin values obtained from the minuted oral glucose tolerance curve at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: pmol*h/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
pmol*h/L | 45016 (22147) | 119704 (46872)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.175, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

21. Secondary Outcome: Glucose at Minute 30 at Week 12.
Description: The glucose at minute 30 is going to be evaluated at week 12 during a minuted oral glucose tolerance curve
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 10.5 (2.0) | 10.0 (1.3)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.392, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.123, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Glucose at Minute 60 at Week 12.
Description: The glucose at minute 60 is going to be evaluated at week 12 during a minuted oral glucose tolerance curve
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 11.1 (3.1) | 11.4 (1.6)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.176, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.268, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

23. Secondary Outcome: Glucose at Minute 90 at Week 12.
Description: The glucose at minute 90 is going to be evaluated at week 12 during a minuted oral glucose tolerance curve
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 9.8 (3.5) | 9.9 (2.3)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.064, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.462, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

24. Secondary Outcome: Glucose at Minute 120 at Week 12.
Description: The glucose at minute 120 is going to be evaluated at week 12 during a minuted oral glucose tolerance curve
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 8.5 (2.1) | 8.8 (2.2)
Statistical Analysis 1: Comparison: Dapagliflozin; Analysis between before and after the intervention; Test type: Superiority; p = 0.346, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Analysis between before and after the intervention; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 12 weeks of the study
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=12) | Placebo (N=12)
Urinary infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes